CLINICAL TRIAL: NCT02754817
Title: A European Multi-centre, Retrospective, Non-interventional Study of the Effectiveness of Xultophy® (Insulin Degludec/Liraglutide) in an Adult Real-world Population With Type 2 Diabetes Mellitus
Brief Title: A Study of the Effectiveness of Xultophy® (Insulin Degludec/Liraglutide) in an Adult Real-world Population With Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9068-4264; U1111-1176-6538 (Other: WHO)
Record Dates: First submitted 2016-04-27; First posted 2016-04-28 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Insulin degludec/liraglutide
  Interventions: Drug: insulin degludec/liraglutide

INTERVENTIONS:
Drug: insulin degludec/liraglutide — This is a non-interventional, chart review study and the patients are treated according to current clinical practice and local licenses upon the treating physicians' decision.

SUMMARY:
This study is conducted in Europe. The aim of the study is to investigate the effectiveness of Xultophy® (insulin degludec/liraglutide) in an adult real-world population with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent obtained before any study-related activities (study-related activities are any procedure related to extraction of data according to the protocol)
* Male or female patients at least 18 years of age at time of informed consent
* Diagnosis of T2DM (type 2 diabetes mellitus)
* Xultophy® initiation prescribed at least 6 months before inclusion in this study (i.e., date of signed informed consent). Patients may or may not be continuing Xultophy® at study inclusion
* Minimum available data:a.) At the time of Xultophy® prescription: HbA1c value (or if unavailable, the most recent HbA1c value within 6 months before the first Xultophy® prescription);b.) At 6 months plus/minus 45 days after first Xultophy® prescription: HbA1c value

Exclusion Criteria:

* Type 1 diabetes
* Previous participation in this study. Participation is defined as having provided informed consent
* Participation in a clinical trial within 6 months before or 12 months after the first Xultophy® prescription (Participation in a non-interventional study is not an exclusion criteria)
* Mental incapacity, unwillingness or inability to provide informed consent, or language barriers precluding adequate understanding or co-operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adults with T2DM. Collecting data reported in medical records of patients with T2DM who received their first prescription of Xultophy® at least 6 months prior to inclusion in this study, no matter whether Xultophy® was continued afterwards.
Sampling Method: Non-Probability Sample
Enrollment: 611 (Actual)
Dates: Start 2016-04-26 (Actual); Primary Completion 2016-10-20 (Actual); Study Completion 2016-10-20 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c (Hemoglobin A1c) | week 0, week 26

SECONDARY OUTCOMES:
Change in HbA1c | Month 0, month 3, month 9, months 12
Percentage of responders for HbA1c below 7 percent (53 mmol/mol) | At 3, 6, 9 and 12 months
Percentage of responders for HbA1c below 7 percent (53 mmol/mol) with no weight gain | At 3, 6, 9 and 12 months
Percentage of responders for HbA1c below 7 percent (53 mmol/mol) with no hypoglycaemic episodes | At 3, 6, 9 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (5):
- Novo Nordisk Investigational Site, Vienna, Austria
- Novo Nordisk Investigational Site, Leipzig, Germany
- Novo Nordisk Investigational Site, Stockholm, Sweden
- Novo Nordisk Investigational Site, Sankt Gallen, Switzerland
- Novo Nordisk Investigational Site, Stevenage, United Kingdom

REFERENCES:
- [Result] Price H, Bluher M, Prager R, Phan TM, Thorsted BL, Schultes B; EXTRA study group. Use and effectiveness of a fixed-ratio combination of insulin degludec/liraglutide (IDegLira) in a real-world population with type 2 diabetes: Results from a European, multicentre, retrospective chart review study. Diabetes Obes Metab. 2018 Apr;20(4):954-962. doi: 10.1111/dom.13182. Epub 2018 Jan 11. PMID 29205856
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com